CLINICAL TRIAL: NCT06492200
Title: Einfluss Ballaststoffreicher Ernährung Auf Das Mikrobiom Und Die Krankheitsaktivität Von Patientinnen Und Patienten Mit Rheumatoider Arthritis
Brief Title: Impact of a High-fiber Diet on the Microbiome and Disease Activity in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: RheinNatur Food GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wuerzburg University Hospital
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Psyllium husks
- Control Group (No Intervention)

INTERVENTIONS:
Other: Psyllium husks — Patients in the intervention group will receive nutritional counseling and will be asked to take 10g (one tablespoon) of ground psyllium husks daily to significantly increase the fiber content of their diet.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if increasing dietary fiber can improve the gut microbiome and reduce disease activity in adults with rheumatoid arthritis (RA). The main questions it aims to answer are:

* Can a higher fiber diet improve gut bacteria and produce beneficial short-chain fatty acids (SCFAs)?
* Does a higher fiber diet reduce RA symptoms and help with weight loss?

Researchers will compare two groups: one group will receive dietary counseling and take 10 grams of psyllium husk daily, while the other group will continue their usual diet.

Participants will:

* Complete dietary questionnaires at the start, 6 months, and 12 months.
* Provide stool samples for gut bacteria and SCFA analysis.
* Have their RA activity and body weight monitored regularly.
* Receive regular phone calls to support the dietary changes.

The study will involve adults with diagnosed RA who can provide informed consent and meet other inclusion criteria.

DETAILED DESCRIPTION:
Background and Rationale:

Rheumatoid arthritis (RA) is an autoimmune disease characterized by chronic inflammation of the joints. Emerging evidence indicates that the gut microbiome plays a crucial role in immune system modulation and may influence the development and progression of RA. Dietary fibers are known to enhance the production of short-chain fatty acids (SCFAs) by gut bacteria, which in turn can have beneficial effects on the immune system. Studies have shown that SCFAs can prevent the onset of RA in animal models and reduce disease activity in humans at risk. Additionally, a fiber-rich diet has been associated with weight loss, which is beneficial for RA patients as lower body weight is linked to reduced disease activity. Despite recommendations from the German Society for Nutrition to consume 30 grams of dietary fiber daily, most individuals fail to meet this target.

Study Objectives and Hypotheses:

The primary objectives of this study are to:

1. Investigate the gut microbiome of patients with established RA and its relationship with disease activity and body weight.
2. Assess whether increasing dietary fiber intake can favorably modify the gut microbiome and increase SCFA production.
3. Determine the impact of a fiber-rich diet on RA disease activity and body weight over a 12-month period.

   The study hypothesizes that a diet higher in dietary fiber will lead to:
   * Improved gut microbiome composition with increased SCFA production.
   * Reduced RA disease activity as measured by DAS28 and CRP.
   * Decreased body weight in overweight RA patients.

   Study Design:

   This is a randomized, controlled, parallel-group clinical trial conducted at the Rheumatology Clinic of the University Clinic Würzburg (UKW). Participants will be randomized into two groups: an intervention group receiving dietary counseling and psyllium husk supplementation, and a control group continuing their usual diet.

   Study Procedures:

   Recruitment:

   - Adult RA patients will be recruited from the Rheumaambulanz at UKW.
   * Inclusion criteria: age >18 years, diagnosis of RA according to the 2010 American College of Rheumatology (ACR) criteria, ability to consent.
   * Exclusion criteria: age <18, lack of consent ability, insufficient German language skills, chronic inflammatory bowel disease, liver cirrhosis, history of mechanical ileus, altered gastrointestinal passage, recent antibiotic use, and recent use of psyllium husk.

   Interventions:

   - Intervention Group: Participants will receive dietary counseling to increase fiber intake and will be asked to consume 10 grams of psyllium husk daily. Regular phone calls will be made to support compliance.

   - Control Group: Participants will maintain their usual diet without additional fiber supplementation.

   Data Collection:
   * Dietary Habits: Questionnaires will be administered at baseline, 6 months, and 12 months to assess dietary fiber intake, protein content, and fat consumption.
   * Body Weight: Participants will be weighed at baseline, 6 months, and 12 months.
   * Disease Activity: DAS28 and CRP levels will be measured at baseline, 6 months, and 12 months.
   * Stool Samples: Collected at baseline, 6 months, and 12 months for microbiome analysis and SCFA quantification.
   * Blood Samples: Routine blood tests including CRP, erythrocyte sedimentation rate (ESR), and metabolic parameters will be evaluated.

   Laboratory Analysis:

   - Stool samples will be analyzed for microbial composition and SCFA content at the Hepatology Laboratory, University Clinic Würzburg. Samples will be stored and destroyed after 10 years.

   - Blood samples will be assessed for routine clinical parameters and lymphocyte characterization.

   Data Analysis:

   - The primary endpoint is the difference in DAS28-CRP scores between the intervention and control groups at 12 months.

   - Statistical tests include Mann-Whitney U for non-parametric data and Fisher's exact test for categorical variables.
   * A sample size of 52 participants (26 per group) is calculated to detect a significant difference with 90% power, accounting for a 20% dropout rate.
   * Multivariate regression analysis will be used to control for potential confounders.

   Quality Assurance:

   - Data will be collected and stored in compliance with General Data Protection Regulation (GDPR) regulations.

   - Data will be pseudonymized for statistical analysis and anonymized for publication.

   - Regular monitoring and auditing will ensure data accuracy and protocol adherence.

   Ethics and Consent:

   - The study protocol, patient information, and consent forms will be reviewed and approved by the local ethics committee at the University Clinic Würzburg.
   * Participation is voluntary, and participants can withdraw at any time without any impact on their standard medical care.

   Publication:

   - Results will be published in peer-reviewed scientific journals in an anonymized format.

   Sponsorship:

   - The study is supported by RheinNatur Food GmbH, which provides the psyllium husk for the intervention.

   This study aims to provide valuable insights into the potential benefits of a high-fiber diet for RA patients, contributing to improved management strategies and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosis of Rheumatoid Arthritis according to the ACR criteria of 2010
* The patient can understand the scope of the study and consents in writing to participate.

Exclusion Criteria:

* Age under 18
* Lack of consent capability
* Insufficient knowledge of the German language
* Chronic inflammatory bowel disease
* Liver cirrhosis
* History of mechanical ileus
* Patients with altered gastrointestinal passage (e.g., stoma patients)
* Use of antibiotics within the past three months
* Use of ground psyllium husks four weeks prior to study inclusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Score 28 (DAS28) | Measurements will be assessed at baseline, 6 months, and 12 months.
  The Disease Activity Score 28 (DAS28) is a composite measure used to assess the activity of rheumatoid arthritis (RA). It is calculated using the number of tender and swollen joints (out of 28 specified joints) and the patient's global health assessment. The DAS28 score ranges from 0 to 9.4, with higher scores indicating higher disease activity. This measure is widely used in clinical practice and research to monitor and evaluate the effectiveness of RA treatments.
C-Reactive Protein (CRP) Level | Measurements will be assessed at baseline, 6 months, and 12 months.
  C-reactive protein (CRP) level is a biomarker used to measure inflammation in the body. Elevated CRP levels are indicative of inflammation and are commonly seen in rheumatoid arthritis patients. CRP levels will be measured using blood tests to assess the inflammatory status of the participants.
Short-Chain Fatty Acids (SCFA) Levels in Stool | Measurements will be assessed at baseline, 6 months, and 12 months.
  The concentration of short-chain fatty acids (SCFAs) in stool samples will be measured. SCFAs, such as acetate, propionate, and butyrate, are produced by the gut microbiota through the fermentation of dietary fibers. These compounds play a crucial role in maintaining gut health and modulating the immune system. The levels of SCFAs will be analyzed to determine the impact of increased dietary fiber intake on gut microbiota composition and function.
Body Weight | Measurements will be assessed at baseline, 6 months, and 12 months.
  Participants' body weight will be measured to assess changes over the study period. Weight measurements will be taken using a standardized and calibrated scale. Changes in body weight will help determine the effect of increased dietary fiber intake on weight management in individuals with rheumatoid arthritis.

SECONDARY OUTCOMES:
Patient Global Assessment of Disease Activity | Measurements will be assessed at baseline, 6 months, and 12 months.
  The Patient Global Assessment of Disease Activity is a subjective measure where participants rate their overall disease activity on a scale from 0 (no disease activity) to 10 (maximum disease activity). This assessment provides insight into the patient's perception of their rheumatoid arthritis and its impact on their daily life.
Health Assessment Questionnaire-Disability Index (HAQ-DI) | Measurements will be assessed at baseline, 6 months, and 12 months.
  The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a self-reported questionnaire used to assess the degree of difficulty a person has in performing daily activities due to their rheumatoid arthritis. The HAQ-DI scores range from 0 (no disability) to 3 (severe disability).
Erythrocyte Sedimentation Rate (ESR) | Measurements will be assessed at baseline, 6 months, and 12 months.
  The Erythrocyte Sedimentation Rate (ESR) is a blood test that measures how quickly erythrocytes (red blood cells) settle at the bottom of a test tube. A faster-than-normal rate may indicate inflammation in the body, which is common in rheumatoid arthritis. ESR levels will be measured to evaluate the inflammatory status of the participants.
Changes in Gut Microbiome Composition | Measurements will be assessed at baseline, 6 months, and 12 months.
  The composition of the gut microbiome will be analyzed using stool samples. This analysis will focus on identifying the types and quantities of bacteria present in the gut. Changes in microbiome composition will be assessed to understand the impact of increased dietary fiber intake on gut health and its potential relationship with rheumatoid arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Schwaneck, M.D., Principal Investigator — University Wuerzburg; Monika Rau, M.D., Study Chair — University Wuerzburg; Michael Gernert, M.D., Study Chair — University Wuerzburg
Locations (1):
- University Würzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No